CLINICAL TRIAL: NCT03315598
Title: Evaluation of an Effectiveness and Safety of the Electroacupuncture in the Management of Intractable Neuropathic Pain: An Open-labeled, Single-arm, Exploratory Pilot Study
Brief Title: Evaluation of an Effectiveness and Safety of the Electroacupuncture in the Management of Intractable Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate professor, Seoul National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1703-024-836
Record Dates: First submitted 2017-10-12; First posted 2017-10-20 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Neuralgia; Neuralgia; Postherpetic; Diabetic Neuropathy, Painful; Failed Back Surgery Syndrome
Keywords: Neuralgia, Acupuncture Treatment
MeSH Terms: conditions — Neuralgia; Neuralgia, Postherpetic; Diabetic Neuropathies; Failed Back Surgery Syndrome | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An open-labeled, single-arm, exploratory pilot study (Experimental): Electroacupunture for 2months
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — lectroacupuncture is a form of acupuncture where a small electric current is passed between pairs of acupuncture needles. According to some acupuncturists, this practice augments the use of regular acupuncture, can restore health and well-being, and is particularly good for treating pain.

SUMMARY:
The investigators will evaluate the effectiveness and safety of acupuncture treatment in refractory neuropathic pain patients.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effectiveness of acupuncture treatment in the patients with the following neuropathic pain related syndrome.

* Postherpetic neuralgia
* Failed back surgery syndrome
* Diabetic neuropathy
* other peripheral neuropathy

Patients with refractory neuropathic pain who do not respond to conservative treatment for more than 3 months should be included. Acupuncture treatment is maintained for 2 months in oriental medicine hospital. The effect is evaluated through the numeric rating score and the validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can adequately write a reportable questionnaire
* Patients who have been diagnosed with one of the following neuropathic pain disease (postherpetic neuralgia, failed back surgery syndrome, diabetic neuropathy, other peripheral neuropathy)
* Patients who failed conservative treatment at Seoul National University Hospital for more than 3 months.
* Patients with NRS 5 points or more
* Patients with painDETECT score 19 points or more

Exclusion Criteria:

* Patients with major mental illness
* Patients with unstable medical conditions
* Pregnant
* Patients who received acupuncture treatment at the site within the past month
* Patients with bleeding tendency
* Patients taking immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline Numeric rating scale pain score (0-10) at 4 weeks | At 4-week follow-up visit
  The Numeric Rating Scale (NRS) is an 11-point scale from 0 to 10 for patient self-reporting of pain. Change from the baseline NRS pain score at 4 weeks will be noted as percentage (%).
Change from baseline Numeric rating scale pain score (0-10) at 8 weeks | At 8-week follow-up visit
  The Numeric Rating Scale (NRS) is an 11-point scale from 0 to 10 for patient self-reporting of pain. Change from the baseline NRS pain score at 4 weeks will be noted as percentage (%).

SECONDARY OUTCOMES:
Change from the score of the short-form McGill Pain Questionnaire at 8 weeks | At 8-week follow-up visit
  The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The SF-MPQ also includes the Present Pain Intensity (PPI) index of the standard MPQ and a visual analogue scale (VAS).
Change from baseline score of Brief Pain Inventory Short Form (BFI-SF) at 8 weeks | At 8-week follow-up visit
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning.
Patients' Global Impression of Change (PGIC) scale | At 8-week follow-up visit
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment.
  1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
5-pointed patient satisfaction scale | At 8-week follow-up visit
  The 5-pointed patient satisfaction scale is an 5-point scale for patient self-reporting of satisfaction with treatment.
  1. Very satisfied
  2. Satisfied
  3. Neither satisfied nor dissatisfied
  4. Dissatisfied
  5. Very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee S, Lee CS, Moon JY, Song HG, Yoo Y, Kim J, Seo H, Lee SH. Electroacupuncture May Improve Burning and Electric Shock-Like Neuropathic Pain: A Prospective Exploratory Pilot Study. J Altern Complement Med. 2020 Dec;26(12):1136-1143. doi: 10.1089/acm.2020.0307. Epub 2020 Oct 19. PMID 33074703